CLINICAL TRIAL: NCT04445155
Title: Modification and Evaluation of the DECIDE Intervention to Improve Parent-provider Interactions in Low-income Parents of Adolescents With Disruptive Impulse Control, and Conduct Disorder
Brief Title: The DECIDE Parent-Provider Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Smith College (Other); University of South Florida (Other); National Institutes of Health (NIH) (NIH); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Ukamaka Marian Oruche, Project Director, Indiana University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1911897011; 5R21MD015150-02 (NIH)
Record Dates: First submitted 2020-02-02; First posted 2020-06-24 (Actual); Results first posted 2024-03-28 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Modified DECIDE Intervention; Treatment as Usual Care Group

STUDY DESIGN:
Intervention Model Description: For clarity, each intervention group was separate and not comparable to other intervention groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Modified DECIDE-Provider Arm (Experimental): 2-4 hour workshop for providers to improve perspective-taking, reduce attributional errors, and increase receptivity to parent participation.
  Interventions: Behavioral: Modified DECIDE Parent and Provider Intervention
- Modified DECIDE-Parent Arm (Experimental): Up to three parent training sessions designed to help patients effectively ask questions and participate in decisions about care.
  Interventions: Behavioral: Modified DECIDE Parent and Provider Intervention
- Provider Subgroup Study (Other): To boost provider recruitment, we sought recommendations from a subgroup of providers. We gave each provider access to the DECIDE online training and the pre- and post-survey.
  Interventions: Behavioral: Modified DECIDE Parent and Provider Intervention
- Treatment as Usual (No Intervention): Control arm

INTERVENTIONS:
Behavioral: Modified DECIDE Parent and Provider Intervention — The parent component will include up to three 60 minutes sessions. Session 1 (Decisions and Agency) is designed to increase awareness of their role in clinical interactions and encourage participation and decision making in care. Session 2 (the Who, How, and Why of Decisions) teach skills for understanding treatment decisions in terms of roles, processes, and reasons involved. Session 3 (Self-efficacy and Consolidation) encourages parents to ask questions about their adolescents' behavioral health and health care and treatment options. The provider component is designed to improve provider communication in three key areas: 1) perspective taking to understand circumstances and perceptions; 2) attributional errors or attributing negative parent behaviors to character traits; and 3) receptivity to parent participation and collaboration.
  Arms: Modified DECIDE-Parent Arm; Modified DECIDE-Provider Arm; Provider Subgroup Study

SUMMARY:
The DECIDE Parent-Provider Intervention is designed to support parents caring for adolescents who are receiving treatment for Disruptive, Impulse-Control, and Conduct disorders. Participating in DECIDE study may help you effectively ask questions and participate in decisions about your adolescent's care. There were three active study arms, each arm had a pre-post design of the DECIDE modified intervention.

DETAILED DESCRIPTION:
Interventions to optimize parent-provider interactions are urgently needed to ensure adolescents aged 3 to 17 years with Disruptive, Impulse-Control, and Conduct disorders (DIC) receive the behavioral health care they need. For these adolescents, behavioral health care is complex, long-term, and requires parental participation. Research shows providers have biases and limited skills and confidence to communicate with these parents to encourage them to voice their concerns and care preferences. Low income and minority parents are at greatest risk of not being involved in their adolescents' behavioral health care, having poor interactions with providers, and are more likely to perceive poor quality of their adolescents' behavioral health care, and low treatment engagement. If unaddressed, poor parent-provider interactions interfere with adolescents' retention in behavioral health care.

No evidence-based interventions have targeted both parents and providers to optimize their interactions and improve behavioral health care for adolescents with DIC. To address these problems, the investigators propose modifying the evidence-based DECIDE intervention to target parents and providers of adolescents with DIC. DECIDE stands for Decide the problem; Explore the questions; Closed or open-ended questions; Identify the who, why, or how of the problem; Direct questions to your health care professional; Enjoy a shared solution. DECIDE was developed for ethnically/racially diverse adult patients with serious mental illness and the latest evidence-based iterations include intervention components targeted to and shown to increase patient activation, provider communication, and patient-provider interactions.

DECIDE has two primary components: 1) three patient training sessions designed to help patients effectively ask questions and participate in decisions about their care: and 2) a 4-hour workshop for providers to improve perspective-taking, reduce attributional errors, and increase receptivity to parent participation and collaboration. The purposes of this two-phase study are: Phase I, Aim 1.

Modify the DECIDE intervention for parents and providers of adolescents with DIC. Phase II, Aim 2. Evaluate the feasibility and acceptability of modified DECIDE. Aim 3. Estimate preliminary effects of modified DECIDE to improve parent, provider, and adolescent outcomes.

Innovative features of this study are the proposed focus on both parents and providers; and inclusion of parent activation and provider communication, which are new in field of child and adolescent behavioral health care, and focus on low income and minority parents. The investigators expect to find that compared to usual care: Hypothesis 3.1. Modified DECIDE parents will show greater improvements in: 1) activation; 2) parent-provider interactions; 3) perceived management of adolescents' behavioral health care, 4) perceived quality of adolescents' behavioral health care, and 5) engagement in adolescents' behavioral healthcare. Hypothesis 3.2. Modified DECIDE providers will show greater improvements in: 1) communication skills; and 2) parent-provider interactions. Hypothesis 3.3. Adolescents of modified DECIDE parents and providers will show higher rates of retention in behavioral health care. Sample will include 16 providers and their parents ( ~ 5 parents per provider, n= 80) recruited from the Child and Adolescents Program of a large safety net health system setting that serves predominately low income and minority persons. Feasibility will be assessed using tracking logs and field notes, and acceptability through parent and provider satisfaction scores and in depth, semi structured interviews. Outcomes will be assessed at baseline and within 4 weeks post- intervention using standardized questionnaires or surveys from parents, providers, and independent observers reports. Effects sizes will be estimated using linear mixed models. If study findings are positive, we will be poised to test the modified DECIDE intervention in a fully powered R01 level randomized, controlled, multi-site clinical trial.

ELIGIBILITY:
Phase 1, Aim 1.

Inclusion Criteria (for Parent Advisory Board; to assist with intervention development):

1. Parents of adolescents with DIC, who are receiving services at Midtown Child and Adolescent Program or CAP. (We will invite parents 1) from our previous study advisory board (n=3), and two who participated in preliminary study 2 that agreed to be contacted for future studies.)

Inclusion Criteria (for Provider Advisory Board; to assist with intervention development):

1. CAP staffs who do not meet the inclusion criteria in phase 2 (i.e. manager and clinical coordinators or supervisors, clinic nurse, advanced practice registered nurses, or psychiatrists). (We will invite two other direct care providers who work in the healthcare system but not at recruitment site. No providers or parents will be excluded on basis of race/ethnicity, gender, or sexual orientation.)

Phase II, Aims 2 and 3.

Inclusion Criteria:

Inclusion Criteria for providers and interns: Providers will be regular paid staff members who are:

1. Associate's or bachelor's or PhD prepared providers who work with parents OR
2. Masters-prepared clinical social workers or mental health counselors and
3. Provide behavioral health services to adolescents and their parents. OR
4. Doctoral level interns (e.g. in psychology) and
5. Provide behavioral health services to adolescents and their parents OR
6. Providers who are bachelor's prepared interns must:

(1) be currently working with a center or private practice to complete requirements for their Master's degree and (2) be providing behavioral health services to adolescents and their parents.

Inclusion Criteria for Guardians: Guardians will have a child or adolescent with DIC receiving services from a participating mental health provider. Parents/guardians meeting all the following criteria are eligible:

1. are aged 21 or older
2. speak English
3. are the guardian (biological parent, adoptive parent, step parent, foster parent, or legal guardian) of the child or adolescent or a parent surrogate serving in a primary caregiver role (referred to as "parents"; if foster parent or legal guardian, ).
4. must have a child or adolescent aged 3 to 17 years with a diagnosis of Disruptive Impulse Control and Conduct Disorder (DIC) by a mental health professional. (This includes children with behavior problems, such as Oppositional Defiant disorder, Conduct disorders, or Intermittent Explosive disorders).
5. Attends regular appointments with a provider
6. Foster parents will be included if they have a child with DIC now or in the past, and regardless of whether that child is receiving services from a participating mental health provider or not.

Exclusion Criteria for parents:

* Show significant cognitive impairment or acute emotional distress on screening
* Have an incarcerated adolescent

No providers or parents will be excluded on basis of race/ethnicity, gender, or sexual orientation.

Specifically for semi-structured interview post intervention. Include: All intervention providers (n = 8) and two of each of their parents (n = 16). To explore different levels of acceptability by parents, for each provider, one parent will be chosen who has a high score (> 3) on the CSQ and one parent who has a low score (< 3). Both parents and providers will be asked about their experience with the intervention, what was helpful or not, and how they would change the intervention.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ukamaka M Oruche, PhD, Principal Investigator — IU Nursing
Locations (5):
- United States (5):
  - Centerstone, Sarasota, Florida
  - Centerstone, Bloomington, Indiana
  - Bowen Center, Fort Wayne, Indiana
  - Sandra Eskenazi Mental Health Center, Indianapolis, Indiana
  - Centerstone, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment as Usual: Control arm: Usual Care
Period: Overall Study
Arm/Group | Modified DECIDE-Provider Arm | Modified DECIDE-Parent Arm | Provider Subgroup Study | Treatment as Usual
Started | 68 | 5 | 16 | 0
Completed | 33 | 3 | 13 | 0
Not Completed | 35 | 2 | 3 | 0
Not completed — Lost to Follow-up | 11 | 2 | 3 | 0
Not completed — Withdrawal by Subject | 8 | 0 | 0 | 0
Not completed — Unable to recruit parent participants so unable to begin study as initially designed | 12 | 0 | 0 | 0
Not completed — Only completed a portion of the final outcome measures (T2) | 4 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: There were no participants enrolled in the Treatment as Usual (Control) Arm. For the Provider Arm, we are only including demographics for those that completed at least one baseline or post-test outcome measure.
Groups:
- Total: Total of all reporting groups
Arm/Group | Modified DECIDE-Provider Arm | Modified DECIDE-Parent Arm | Provider Subgroup Study | Treatment as Usual | Total
Number analyzed (Participants) | 53 | 5 | 16 | 0 | 74
Age, Categorical [Count of Participants; unit: Participants] — Population: For Provider Arm, two participants did not report their age. For Parent Arm, two participants did not report their age. Age was not collected for the Provider Subgroup Arm.
  Participants
    number analyzed (Participants) | 51 | 3 | 0 | 0 | 54
    <=18 years | 0 | 0 |  |  | 0
    Between 18 and 65 years | 50 | 3 |  |  | 53
    >=65 years | 1 | 0 |  |  | 1
Age, Continuous [Median (Full Range); unit: years] — Population: For the Provider Arm, two participants did not report their age. For Parent Arm, two participants did not report their age. Age was not collected for the Provider Subgroup Arm.
  years
    number analyzed (Participants) | 51 | 3 | 0 | 0 | 54
    (all) | 33 [22 to 66] | 47 [43 to 55] |  |  | 34 [22 to 66]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: For the Provider Arm, 2 participants did not report sex. Sex was not collected for the Provider Subgroup Arm.
  Participants
    number analyzed (Participants) | 51 | 5 | 0 | 0 | 56
    Female | 48 | 4 |  |  | 52
    Male | 3 | 1 |  |  | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Ethnicity was not collected for the Provider Subgroup Arm.
  Participants
    number analyzed (Participants) | 53 | 5 | 0 | 0 | 58
    Hispanic or Latino | 2 | 0 |  |  | 2
    Not Hispanic or Latino | 49 | 5 |  |  | 54
    Unknown or Not Reported | 2 | 0 |  |  | 2
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Race was not collected for the Provider Subgroup Arm.
  Participants
    number analyzed (Participants) | 53 | 5 | 0 | 0 | 58
    American Indian or Alaska Native | 0 | 0 |  |  | 0
    Asian | 1 | 0 |  |  | 1
    Native Hawaiian or Other Pacific Islander | 0 | 0 |  |  | 0
    Black or African American | 7 | 1 |  |  | 8
    White | 39 | 4 |  |  | 43
    More than one race | 2 | 0 |  |  | 2
    Unknown or Not Reported | 4 | 0 |  |  | 4
Region of Enrollment [Number; unit: participants]
  United States | 53 | 5 | 16 |  | 74
Parent Needs & Resources Domain of CANS - Provider Arm Only [Median (Inter-Quartile Range); unit: units on a scale] — Parent Needs & Resources Domain of CANS is measured using three items from the Parent Needs & Resources Domain of the Child and Adolescent Needs and Strengths (CANS), Involvement with Care, Knowledge, and Organization. Each item is scored 0, 1, 2, or 3. A domain score is created by calculating the sum of the items. The domain score ranges from 0 to 9 with higher scores meaning more need/less strength. Population: In the Provider Arm, one participant did not complete this scale at baseline. This scale was not collected in the other study arms.
  units on a scale
    number analyzed (Participants) | 52 | 0 | 0 | 0 | 52
    (all) | 3.5 [3 to 5] |  |  |  | 3.5 [3 to 5]
Parent Activation Measure Mental Health (P-PAM-MH) - Parent Arm Only [Median (Inter-Quartile Range); unit: units on a scale] — Parent Activation Measure Mental Health is measured using a 13-item scale. Items are scored using a 4-point Likert-type scale (1 = disagree strongly to 4 = agree strongly). Raw item scores are summed and scaled from 0-100. Higher scores indicate greater activation. Population: This scale was only collected in the Parent Arm.
  units on a scale
    number analyzed (Participants) | 0 | 5 | 0 | 0 | 5
    (all) |  | 43.1 [39.2 to 51.0] |  |  | 43.1 [39.2 to 51.0]
Parent Participation Engagement Measure (PPEM) - Provider and Parent Arm Only [Mean (Standard Deviation); unit: units on a scale] — Parent Participation Engagement Measure is measured using a 5-item scale that measures the frequency with which the parent engaged during clinical encounter or parent-provider interaction. Behaviors assessed include asking questions, making suggestions or sharing one's opinion or point of view, and participating in therapeutic activities. Response options are on a 5-point scale ranging from 1 = "not at all" to 5 = "very much". A mean score is calculated using all 5 items and has a range of 1 to 5. Higher scores indicate greater frequency of parent engagement. Population: In the Provider Arm, one participant did not complete this scale at baseline. This scale was only collected in the Provider Arm and Parent Arm.
  units on a scale
    number analyzed (Participants) | 52 | 5 | 0 | 0 | 57
    (all) | 3.1 (0.9) | 2.6 (1.7) |  |  | 3.1 (1.0)
Familiarity with Perspective Taking - Provider Arm and Provider Subgroup Arm Only [Count of Participants; unit: Participants] — Familiarity with perspective taking is measured using a single item that measures familiarity with concept of perspective taking. The response options are 0=Not at all, 1=A little bit, and 2=A lot. A higher score means more familiarity with the concept of perspective taking. Population: In the Provider Arm, one participant did not complete this scale at baseline. This scale was only collected in the Provider Arm and Provider Subgroup Arm.
  Participants
    number analyzed (Participants) | 52 | 0 | 16 | 0 | 68
    1 = Not at all | 6 |  | 5 |  | 11
    2 = A little bit | 22 |  | 5 |  | 27
    3 = A lot | 24 |  | 6 |  | 30
Familiarity with Attribution Errors - Provider Arm and Provider Subgroup Arm Only [Count of Participants; unit: Participants] — Familiarity with attribution errors is measured using a single item that measures familiarity with concept of attribution errors. The response options are 1=Not at all, 2=A little bit, and 3=A lot. A higher score means more familiarity with the concept of attribution errors. Population: In the Provider Arm, one participant did not complete this scale at baseline. This scale was only collected in the Provider Arm and Provider Subgroup Arm.
  Participants
    number analyzed (Participants) | 52 | 0 | 16 | 0 | 68
    1 = Not at all | 17 |  | 6 |  | 23
    2= A little | 25 |  | 8 |  | 33
    3 = A lot | 10 |  | 2 |  | 12
Familiarity with Receptivity - Provider Arm and Provider Subgroup Arm Only [Count of Participants; unit: Participants] — Familiarity with receptivity is measured using a single item that measures familiarity with concept of receptivity. The response options are 1=Not at all, 2=A little bit, and 3=A lot. A higher score means more familiarity with the concept of receptivity. Population: In the Provider Arm, two participants did not complete this scale at baseline. This scale was only collected in the Provider Arm and Provider Subgroup Arm.
  Participants
    number analyzed (Participants) | 51 | 0 | 16 | 0 | 67
    1 = Not at all | 9 |  | 4 |  | 13
    2 = A little | 28 |  | 5 |  | 33
    3 = A lot | 14 |  | 7 |  | 21
Communication Scale of the Kim Alliance Scale Refined (KAS-R) - Parent Arm Only [Median (Inter-Quartile Range); unit: units on a scale] — Communication scale of the Kim Alliance Scale Refined is measured using a 4-item scale that measures perception of parent-provider communication. Response categories include 1 = never to 4 = always. Items are summed with higher scores indicating higher quality of communication (range = 4 to 16). Population: This scale was only collected in the Parent Arm.
  units on a scale
    number analyzed (Participants) | 0 | 5 | 0 | 0 | 5
    (all) |  | 13 [4 to 14] |  |  | 13 [4 to 14]
Perceived Efficacy in Parent-Physician Interactions (PEPPI)-Short Form - Parent Arm Only [Median (Inter-Quartile Range); unit: units on a scale] — Perceived Efficacy in Parent-Physician Interactions is measured using a 10-item scale that measures patient's confidence in ability to elicit and understand information from and communicate information to providers. Response categories are 1 = low to 10 = high. A total score is obtained by summing all individual scores with higher scores indicating greater perceived confidence in ability to elicit and understand information from and communicate information to providers (range = 10 to 100). Population: This scale was only collected in the Parent Arm.
  units on a scale
    number analyzed (Participants) | 0 | 5 | 0 | 0 | 5
    (all) |  | 30 [19 to 31] |  |  | 30 [19 to 31]
Perception of Care Quality Survey - Parent Arm Only [Median (Inter-Quartile Range); unit: units on a scale] — Perception of Care Quality is measured using a single item that measures overall rating of parent's perception of care quality. Reponses are 1 to 10 where 1=Worst possible care to 10=Best possible care. Higher scores indicate perceptions of higher quality of care. Population: This item was only collected in the Parent Arm.
  units on a scale
    number analyzed (Participants) | 0 | 5 | 0 | 0 | 5
    (all) |  | 7 [5 to 7] |  |  | 7 [5 to 7]

OUTCOME MEASURES:

1. Primary Outcome: Change in Parent Needs & Resources Domain of CANS - Provider Arm Only
Description: Change in Parent Needs & Resources Domain of CANS is measured using three items from the Parent Needs & Resources Domain of the Child and Adolescent Needs and Strengths (CANS), Involvement with Care, Knowledge, and Organization. Each item is scored 0, 1, 2, or 3. A domain score is created by calculating the sum of the items. The domain score ranges from 0 to 9 with higher scores meaning more need/less strength and is calculated at baseline and immediately post-intervention. Change from baseline equals the score immediately post-intervention minus the score at baseline. Changes can range from -9 to 9 with positive values indicating in increase in need/decrease in strength.
Time Frame: baseline and immediately post intervention (T2), up to 4 weeks
Population: In the Provider Arm, 34 participants completed both baseline and immediately post-intervention timepoints. This scale was not collected in the other study arms.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Modified DECIDE-Provider Arm | Modified DECIDE-Parent Arm | Provider Subgroup Study | Treatment as Usual
Number analyzed (Participants) | 34 | 0 | 0 | 0
units on a scale | 0 [-2 to 0] |  |  |
Statistical Analysis 1: Comparison: Modified DECIDE-Provider Arm; Null Hypothesis: The distributions of the scores are the same at baseline and immediately post-intervention. Alternative Hypothesis: The distributions of the scores are different at baseline and immediately post-intervention; Test type: Superiority; p = 0.125, Wilcoxon Signed-Rank test

2. Primary Outcome: Change in Parent Activation Measure Mental Health (P-PAM-MH) - Parent Arm Only
Description: Change in Parent Activation Measure Mental Health is measured using a 13-item scale. Items are scored using a 4-point Likert-type scale (1 = disagree strongly to 4 = agree strongly). Raw item scores are summed and scaled from 0-100. Higher scores indicate greater activation and is calculated at baseline and immediately post-intervention. Change from baseline equals the score immediately post-intervention minus the score at baseline. Changes can range from -100 to 100 with positive values indicating an increase in activation.
Time Frame: baseline and immediately post intervention (T2), up to 4 weeks
Population: In the Parent Arm, 4 participants completed both baseline and immediately post-intervention timepoints. This scale was not collected in the other study arms.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Modified DECIDE-Provider Arm | Modified DECIDE-Parent Arm | Provider Subgroup Study | Treatment as Usual
Number analyzed (Participants) | 0 | 4 | 0 | 0
units on a scale |  | 15.7 [4.9 to 25.5] |  |

3. Secondary Outcome: Change in Parent Participation Engagement Measure (PPEM) - Provider and Parent Arm Only
Description: Change in Parent Participation Engagement Measure is measured using a 5-item scale that measures the frequency with which the parent engaged during clinical encounter or parent-provider interaction. Behaviors assessed include asking questions, making suggestions or sharing one's opinion or point of view, and participating in therapeutic activities. Response options are on a 5-point scale ranging from 1 = "not at all" to 5 = "very much". A mean score is calculated using all 5 items and has a range of 1 to 5. Higher scores indicate greater frequency of parent engagement and is calculated at baseline and immediately post intervention. Change from baseline equals the score immediately post-intervention minus the score at baseline. Changes can range from -4 to 4 with positive values indicating an increase in activation.
Time Frame: baseline and immediately post intervention (T2), up to 4 weeks
Population: In the Provider Arm, 34 participants completed both baseline and immediately post-intervention timepoints. In the Parent Arm, 4 participants completed both baseline and immediately post-intervention timepoints. This scale was not collected in the other study arms.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Modified DECIDE-Provider Arm | Modified DECIDE-Parent Arm | Provider Subgroup Study | Treatment as Usual
Number analyzed (Participants) | 34 | 4 | 0 | 0
units on a scale | 0.4 (0.9) | 0.5 (0.8) |  |
Statistical Analysis 1: Comparison: Modified DECIDE-Provider Arm; Null Hypothesis: The means of the scores are the same at baseline and immediately post-intervention. Alternative Hypothesis: The means of the scores are different at baseline and immediately post-intervention; Test type: Superiority; p = 0.011, Paired t-test

4. Secondary Outcome: Change in Familiarity With Perspective Taking - Provider Arm and Provider Subgroup Arm Only
Description: Change in familiarity with perspective taking is measured using a single item that measures familiarity with concept of perspective taking. The response options are 0=Not at all, 1=A little bit, and 2=A lot. A higher score means more familiarity with the concept of perspective taking and is calculated at baseline and post intervention. Change from baseline equals the score immediately post-intervention minus the score at baseline. Changes can range from -2 to 2 with positive values indicating an increase in familiarity with the concept of perspective taking.
Time Frame: baseline and immediately post intervention (T2), up to 4 weeks
Population: In the Provider Arm, 35 participants completed both baseline and immediately post-intervention timepoints. In the Provider Subgroup Arm, 13 completed both baseline and immediately post-intervention timepoints. This scale was only collected in the Provider Arm and Provider Subgroup Arm.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Modified DECIDE-Provider Arm | Modified DECIDE-Parent Arm | Provider Subgroup Study | Treatment as Usual
Number analyzed (Participants) | 35 | 0 | 13 | 0
units on a scale | 0 [0 to 1] |  | 1 [0 to 1] |
Statistical Analysis 1: Comparison: Modified DECIDE-Provider Arm; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.002, Wilcoxon Signed-Rank test
Statistical Analysis 2: Comparison: Provider Subgroup Study; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.008, Wilcoxon Signed-Rank test

5. Secondary Outcome: Change in Familiarity With Attribution Errors - Provider Arm and Provider Subgroup Arm Only
Description: Change in familiarity with attribution errors is measured using a single item that measures familiarity with concept of attribution errors. The response options are 1=Not at all, 2=A little bit, and 3=A lot. A higher score means more familiarity with the concept of attribution errors and is calculated at baseline and post intervention. Change from baseline equals the score immediately post-intervention minus the score at baseline. Changes can range from -2 to 2 with positive values indicating an increase in familiarity with the concept of attribution errors.
Time Frame: baseline and immediately post intervention (T2), up to 4 weeks
Population: In the Provider Arm, 35 participants completed both baseline and immediately post-intervention timepoints. In the Provider Subgroup Arm, 13 completed both baseline and immediately post-intervention timepoints. This scale was was only collected in the Provider Arm and Provider Subgroup Arm.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Modified DECIDE-Provider Arm | Modified DECIDE-Parent Arm | Provider Subgroup Study | Treatment as Usual
Number analyzed (Participants) | 35 | 0 | 13 | 0
units on a scale | 1 [0 to 1] |  | 1 [1 to 1] |
Statistical Analysis 1: Comparison: Modified DECIDE-Provider Arm; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, Wilcoxon Signed-Rank test
Statistical Analysis 2: Comparison: Provider Subgroup Study; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.002, Wilcoxon Signed-Rank test

6. Secondary Outcome: Change in Familiarity With Receptivity - Provider Arm and Provider Subgroup Arm Only
Description: Change in familiarity with receptivity is measured using a single item that measures familiarity with concept of receptivity. The response options are 1=Not at all, 2=A little bit, and 3=A lot. A higher score means more familiarity with the concept of receptivity and is calculated at baseline and post intervention. Change from baseline equals the score immediately post-intervention minus the score at baseline. Changes can range from -2 to 2 with positive values indicating an increase in familiarity with the concept of receptivity.
Time Frame: baseline and immediately post intervention (T2), up to 4 weeks
Population: In the Provider Arm, 34 participants completed both baseline and immediately post-intervention timepoints. In the Provider Subgroup Arm, 13 completed both baseline and immediately post-intervention timepoints. This scale was only collected in the Provider Arm and Provider Subgroup Arm.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Modified DECIDE-Provider Arm | Modified DECIDE-Parent Arm | Provider Subgroup Study | Treatment as Usual
Number analyzed (Participants) | 35 | 0 | 13 | 0
units on a scale | 0 [0 to 1] |  | 0 [0 to 1] |
Statistical Analysis 1: Comparison: Modified DECIDE-Provider Arm; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, Wilcoxon Signed-Rank test
Statistical Analysis 2: Comparison: Provider Subgroup Study; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.125, Wilcoxon Signed-Rank test

7. Secondary Outcome: Change in Communication Scale of the Kim Alliance Scale Refined (KAS-R): Post-intervention - Parent Arm Only
Description: Change in the Communication scale of the Kim Alliance Scale Refined is measured using a 4-item scale that measures perception of parent-provider communication. Response categories include 1 = never to 4 = always. Items are summed with higher scores indicating higher quality of communication and is calculated at baseline and post intervention (range 4 to 16). Change from baseline equals the score immediately post-intervention minus the score at baseline. Changes can range from -12 to 12 with positive values indicating an increase in quality of communication.
Time Frame: baseline and immediately post intervention (T2), up to 4 weeks
Population: In the Parent Arm, 3 participants completed both baseline and immediately post-intervention timepoints. This scale was not collected in the other study arms.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Modified DECIDE-Provider Arm | Modified DECIDE-Parent Arm | Provider Subgroup Study | Treatment as Usual
Number analyzed (Participants) | 0 | 3 | 0 | 0
units on a scale |  | 0 [0 to 1] |  |

8. Secondary Outcome: Change in Perceived Efficacy in Parent-Physician Interactions (PEPPI)-Short Form: Post-intervention - Parent Arm Only
Description: Change in Perceived Efficacy in Parent-Physician Interactions is measured using a 10-item scale that measures patient's confidence in ability to elicit and understand information from and communicate information to providers. Response categories are 1 = low to 10 = high. A total score is obtained by summing all individual scores with higher scores indicating greater perceived confidence in ability to elicit and understand information from and communicate information to providers (range = 10 to 100). Change from baseline equals the score immediately post-intervention minus the score at baseline. Changes can range from -90 to 90 with positive values indicating an increase confidence in ability to elicit and understand information from and communicate information to providers.
Time Frame: baseline and immediately post intervention (T2), up to 4 weeks
Population: In the Parent Arm, 3 participants completed both baseline and immediately post-intervention timepoints. This scale was only collected in the Parent Arm.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Modified DECIDE-Provider Arm | Modified DECIDE-Parent Arm | Provider Subgroup Study | Treatment as Usual
Number analyzed (Participants) | 0 | 3 | 0 | 0
units on a scale |  | 14 [8 to 15] |  |

9. Secondary Outcome: Change in Perception of Care Quality Survey: Post-intervention - Parent Only
Description: Change in Perception of Care Quality is measured using a single item that measures overall rating of parent's perception of care quality. Reponses are 1 to 10 where 1=Worst possible care to 10=Best possible care. Higher scores indicate perceptions of higher quality of care. Item was collected at baseline and immediately post intervention. Change from baseline equals the score immediately post-intervention minus the score at baseline. Changes can range from -9 to 9 with positive values indicating an increase in rating of perception of higher quality of care.
Time Frame: baseline and immediately post intervention (T2), up to 4 weeks
Population: In the Parent Arm, 3 participants completed both baseline and immediately post-intervention timepoints. This item was only collected in the Parent Arm.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Modified DECIDE-Provider Arm | Modified DECIDE-Parent Arm | Provider Subgroup Study | Treatment as Usual
Number analyzed (Participants) | 0 | 3 | 0 | 0
units on a scale |  | 0 [0 to 3] |  |

ADVERSE EVENTS:
Time Frame: 4 months from baseline
Description: 89 participants at risk for Serious Adverse Events 89 participants at risk for All-Cause Mortality 89 participants at risk for Other (not Including Serious)
Arm/Group | Modified DECIDE-Provider Arm | Modified DECIDE-Parent Arm | Provider Subgroup Study | Treatment as Usual
All-Cause Mortality (participants affected / at risk) | 0/68 | 0/5 | 0/16 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/68 | 0/5 | 0/16 | 0/0
Other Adverse Events (participants affected / at risk) | 0/68 | 0/5 | 0/16 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2022-12-06): https://cdn.clinicaltrials.gov/large-docs/55/NCT04445155/Prot_002.pdf
  • Statistical Analysis Plan (2023-12-13): https://cdn.clinicaltrials.gov/large-docs/55/NCT04445155/SAP_003.pdf
  • Informed Consent Form (2022-12-06): https://cdn.clinicaltrials.gov/large-docs/55/NCT04445155/ICF_004.pdf